CLINICAL TRIAL: NCT03466606
Title: Implementation of a Trimodal Prehabilitation Program as a Preoperative Optimization Strategy in Cardiac Surgery
Brief Title: Implementation of a Trimodal Prehabilitation Program as a Preoperative Optimization Strategy in Cardiac Surgery and Heart Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Graciela Martinez-Palli, Head of Anesthesia Department, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI1700852
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease; Valvular Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Personalized supervised resistance training and program to promote physical activity and healthy lifestyles
  Interventions: Behavioral: pre-habilitation
- Control (No Intervention): Conventional treatment

INTERVENTIONS:
Behavioral: pre-habilitation — Personalized supervised resistance training and program to promote physical activity and healthy lifestyles
  Arms: Prehabilitation

SUMMARY:
Pre-habilitation programs that combine physical training, nutritional support and emotional reinforcement have demonstrated efficacy as presurgical optimization strategies in the context of digestive surgery. The experience in patients at risk for cardiac surgery, one of those associated with higher morbidity and mortality, is anecdotal. Main objective: to evaluate the feasibility, efficacy and cost-effectiveness of a pre-habilitation program for the improvement of preoperative functional capacity in high-risk and intermediate risk groups for cardiac surgery and its impact on the reduction of postoperative complications (primary endpoint). Secondary objectives: (i) in-hospital stay; (ii) symptoms, quality of life, (iii) evaluation of information and communication technologies (ICT) as a support for the pre-habilitation, and (iv) design and validation of indicators for a future large-scale implementation of this type of intervention.

Design: Subproject: #1: Prospective study of the efficacy of prehabilitation in heart transplant candidates during the study period. The results will be compared with historical records; #2: Randomized controlled trial with a 1:1 ratio to assess the efficacy of prehabilitation in patients undergoing elective coronary revascularization or valve replacement surgery. Subjects: Subproject #1: 40 patients candidates for heart transplantation. Subproject #2: 80 patients in the prehabilitation group and 80 controls in which a conventional treatment will be performed. Intervention: (i) personalized supervised resistance training, and (ii) program to promote physical activity and healthy lifestyles. The overall duration of the intervention is estimated to be at least 4-6 weeks (variable in each subproject). The support with ICTs will be a significant aspect of the program in which the adaptation of the personal health folder of Catalonia (Cat@SalutLaMevaSalut) will be fundamental.

ELIGIBILITY:
Inclusion Criteria:

* Subproject #1: Heart transplant candidates
* Subproject #2: Patients awaiting for coronary artery bypass or valve surgery with an expected waiting time for surgery of 8-12 weeks

Exclusion Criteria:

* Dynamic left ventricular outflow tract obstruction (> 40 mmHg)
* Arrythmia induced by exercise
* Emergent surgery
* Unstable cardiac disease
* Unstable severe co-morbid disease
* Disabling orthopedic and neuromuscular disease
* Cognitive impairment
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative complications graded by Clavien Dindo classification. | 30 days or the postoperative hospital stay if longer than 30 days
  The classification's basic principle is to grade complications according to the treatment that is induced to treat the complication. It consists of 5 grades with 2 grades being further subdivided.

SECONDARY OUTCOMES:
Length of stay | 30 days or the postoperative hospital stay if longer than 30 days
  The total length, in days, that patient stays in a hospital after surgery (including the day of the surgery)

OTHER OUTCOMES:
Mortality | 6 months
  Yes or no
Training induced enhancement of aerobic capacity | baseline, after the 4-6 week endurance training program (before surgery)
  Endurance time variation pre- and post intervention
To evaluate de magnitude of cognitive performance change from the preoperative period to 3 months after cardiac surgery | At baseline and 3 months after surgery
  two questions exploring subjective cognitive, and eight tests exploring different cognitive domains (Memory Alteration Test, the digit forwards and backwards from the Wechsler Adult Intelligence Scale, forms A and B from the Trail Making Test, the Symbol Digit Modalities Test, the Semantic Fluency Test, and the Mini-Mental State Examination (MMSE).
To evaluate the incidence of postoperative cognitive disfunction at 3 months after surgery | At 3 months after surgery
  two questions exploring subjective cognitive, and eight tests exploring different cognitive domains (Memory Alteration Test, the digit forwards and backwards from the Wechsler Adult Intelligence Scale, forms A and B from the Trail Making Test, the Symbol Digit Modalities Test, the Semantic Fluency Test and the Mini-Mental State Examination (MMSE).
Health-related quality of life | at baseline and after the 4-6 week endurance training program (before surgery)
  EuroQol-5D, EQ5D questionnaire
Analysis of the barriers for the use of communication and information technologies in prehabilitation program | 6 weeks
  Specific questionnaire, study compliance

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Martinez palli, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinic Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lopez-Hernandez A, Gimeno-Santos E, Navarro-Ripoll R, Arguis MJ, Lopez-Baamonde M, Sanz-de la Garza M, Sandoval E, Castella M, Martinez-Palli G. Multimodal prehabilitation as a strategy to reduce postoperative complications in cardiac surgery: A randomised controlled trial. Eur J Anaesthesiol. 2025 Nov 1;42(11):987-996. doi: 10.1097/EJA.0000000000002236. Epub 2025 Jul 16. PMID 40673713
- [Derived] Lopez-Hernandez A, Gimeno-Santos E, Navarro-Ripoll R, Arguis MJ, Romano-Andrioni B, Lopez-Baamonde M, Teres S, Sanz-de la Garza M, Martinez-Palli G. Differential response to preoperative exercise training in patients candidates to cardiac valve replacement. BMC Anesthesiol. 2024 Aug 9;24(1):280. doi: 10.1186/s12871-024-02671-x. PMID 39123146
- [Derived] Coca-Martinez M, Lopez-Hernandez A, Montane-Muntane M, Arguis MJ, Gimeno-Santos E, Navarro-Ripoll R, Perdomo J, Lopez-Baamonde M, Rios J, Moises J, Sanz de la Garza M, Sandoval E, Romano B, Sebio R, Dana F, Martinez-Palli G. Multimodal prehabilitation as strategy for reduction of postoperative complications after cardiac surgery: a randomised controlled trial protocol. BMJ Open. 2020 Dec 22;10(12):e039885. doi: 10.1136/bmjopen-2020-039885. PMID 33371022

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03466606/Prot_SAP_000.pdf
  • Informed Consent Form: Informed consent form subproject2 general (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03466606/ICF_001.pdf
  • Informed Consent Form: Informed consent form subproject2 intervention (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03466606/ICF_002.pdf
  • Informed Consent Form: Informed consent form subproject1 transplantation (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT03466606/ICF_003.pdf